CLINICAL TRIAL: NCT03694665
Title: Non-invasive Assessment of Lung Recruitment in Morbid Obese Patients Undergoing Bariatric Surgery
Brief Title: Monitoring Lung Recruitment Maneuver in Anesthetized Morbidly Obese
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Privado de Comunidad de Mar del Plata (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HPC-
Record Dates: First submitted 2016-08-01; First posted 2018-10-03 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2018-08

CONDITIONS: Atelectasis
Keywords: airways pressure; mechanical ventilation; Atelectasis
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Morbidly anesthetized obese (Other): Morbidly obese patients undergoing bariatric surgery (single-arm study) will receive a Lung recruitment maneuver to treat atelectasis..
  Interventions: Other: Lung recruitment maneuver

INTERVENTIONS:
Other: Lung recruitment maneuver — A Lung recruitment maneuver is aimed to resolve atelectasis during mechanical ventilation. It consists in a brief and controlled increment in airways pressure using pressure control ventilation. Positive end-expiratory pressure (PEEP) is increases every 5 centimeters of water (cmH2O), from 0 to 20 cmH2O keeping a fixed driving pressure of 20 cmH2O. A final step of 40 cmH2O of plateau pressure was maintained for 10 breaths, returning then to standard ventilatory settings.

SUMMARY:
Morbid obese patients present changes in respiratory physiology caused by weight overload. Intraoperative atelectasis is a pulmonary complication that affects not only gas exchange but also respiratory mechanics. The present study was aimed to test the role of different parameters for monitoring the treatment of atelectasis by a lung recruitment maneuver.

DETAILED DESCRIPTION:
This is a prospective study perform in 30 anesthetized morbidly obese undergoing bariatric surgery. Lung mechanics and volumetric capnography will be non-invasively assessed during laparoscopy. Esophageal pressure will be measured by an esophageal balloon to measure transpulmonary pressure. A lung recruitment maneuver will be done. The optimum level of positive end-expiratory pressure (PEEP) is defined as the PEEP level when transpulmonary pressure remains positive during the PEEP titration trial of the recruitment maneuver. Lung collapse is detected when transpulmonary pressure becomes negative. The behavior of the studied volumetric capnography and lung mechanics parameters will be compared with the reference transpulmonary pressure signal.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) > 40 kg/m2
* Written inform consent
* Scheduled for bariatric surgery
* American Society of Anesthesia physical status II-III

Exclusion Criteria:

* Acute pulmonary disease
* Emergency surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-09-11 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-05-17 (Actual)

PRIMARY OUTCOMES:
Measurement of the optimum positive end-expiratory pressure in anesthetized morbidly obese patients | intraoperative
  Comparison between a reference method (esophageal balloon) with volumetric capnography.

CONTACTS AND LOCATIONS:
Overall Officials: Gerardo Tusman, MD, Principal Investigator — Hospital Privado de Comunidad
Locations (1):
- Hospital Privado de Comunidad, Mar del Plata, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No